CLINICAL TRIAL: NCT05283239
Title: Impact of HPV Integration on the Prognosis of Women With Persistent HR-HPV Infection：a Multi-center Cohort Study in China
Brief Title: Research About Impact of HPV Integration on the Prognosis of Women With Persistent HR-HPV Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Binhua Dong, Principal Investigator, Fujian Maternity and Child Health Hospital
Other Study IDs: HIHP2201
Record Dates: First submitted 2022-02-17; First posted 2022-03-16 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: HPV Infection; LSIL, Low-Grade Squamous Intraepithelial Lesions; HSIL, High-Grade Squamous Intraepithelial Lesions; Virus Integration
MeSH Terms: conditions — Papillomavirus Infections; Squamous Intraepithelial Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples from cervix and vagina containing related cells, tissues and secretions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with persistent HR-HPV infection: In the enrollment, women with persistent HR-HPV infection for more than 18 months will be included in this study. All participants will be followed up at 6th month, 12th month, 18th month and 24th month after baseline of recruitment.
  Interventions: Other: Follow up

INTERVENTIONS:
Other: Follow up — Participants will be followed up at 6th，12th, 18th and 24th months with HPV viral integration/genotyping tests, thinprep cytologic tests (TCT) for cervix and vaginal secretion tests. Colposcopy and biopsy will be conducted for participants if necessary.

SUMMARY:
Clinically, patients with persistent HR-HPV infection for more than 18 months or HR-HPV infection with CIN2 + need regular colposcopic biopsy to assess the outcome and progression of the disease. A total of 1000 participants with persistent HR-HPV infection (100 cases/center) were recruited from multiple centers, and HPV integration status and vaginal flora diversity were sequenced at baseline, 6th month, 12th month and 24th month, respectively, through prospective cohort studies. And to evaluate the influence of HPV integration status and flora changes on the prognosis of women with persistent HR-HPV infection.

DETAILED DESCRIPTION:
This study aims to: 1) determine the association between HPV integration and natural outcome in women with persistent HR-HPV infection. 2) determine the prognostic value of different HPV integration status in women with persistent HR-HPV infection. 3) determine the relationship between the integration status of different HPV genes in the cervix and the diversity of vaginal flora in women with persistent HR-HPV infection, and its prognostic value in women with LSIL and HSIL.

ELIGIBILITY:
Inclusion Criteria:

* Non pregnant people with sexual history；
* Persistent infection of the same type of HR-HPV for more than 18 months or HR-HPV infection with CIN2 +;
* No history of previous surgery at the cervical site.
* Asexual life, no vaginal medication or flushing before 72 hours of sampling.

Exclusion Criteria:

* Within 8 weeks after pregnancy or postpartum.
* Patients with history of genital tract tumor.
* History of HPV vaccination.
* Previous history of hysterectomy, cervical surgery, pelvic radiotherapy Historical.
* In recent one month, she has received genital tract infection, HPV or other STDs treatment related to the infection of mycoplasma.
* Use antibiotics or vaginal microecological improvement products in recent 1 month.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese women with persistent infection of the same type of HR-HPV for more than 18 months or HR-HPV infection with CIN2 +.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cervical histopathology testing at baseline | Baseline
  Cervical histopathology was performed at baseline for all participants.
Cervical histopathology testing at 6-month follow-up | 6-month follow-up
  Cervical histopathology was performed at 6-month follow-up for cervical HR-HPV infection or cytology abnormalities women
Cervical histopathology testing at 12-month follow-up | 12-month follow-up
  Cervical histopathology was performed at 12-month follow-up for cervical HR-HPV infection or cytology abnormalities women
Cervical histopathology testing at 18-month follow-up | 18-month follow-up
  Cervical histopathology was performed at 18-month follow-up for cervical HR-HPV infection or cytology abnormalities women
Cervical histopathology testing at 24-month follow-up | 24-month follow-up
  Cervical histopathology was performed at 24-month follow-up for cervical HR-HPV infection or cytology abnormalities women
Human Papillomavirus (HPV) virus integration test at baseline | Baseline
  Human Papillomavirus (HPV) virus integration test was performed at baseline for all participants.
Human Papillomavirus (HPV) virus integration test at 6-month follow-up | 6-month follow-up
  Human Papillomavirus (HPV) virus integration test was performed at 6-month follow-up for all participants.
Human Papillomavirus (HPV) virus integration test at 12-month follow-up | 12-month follow-up
  Human Papillomavirus (HPV) virus integration test was performed at 12-month follow-up for all participants.
Human Papillomavirus (HPV) virus integration test at 18-month follow-up | 18-month follow-up
  Human Papillomavirus (HPV) virus integration test was performed at 18-month follow-up for all participants.
Human Papillomavirus (HPV) virus integration test at 24-month follow-up | 24-month follow-up
  Human Papillomavirus (HPV) virus integration test was performed at 24-month follow-up for all participants.
Cervical cytology testing at baseline | Baseline
  All participants were tested for cervical cytology at the time of baseline.
Cervical cytology testing at 6-month follow-up | 6-month follow-up
  All participants were tested for Cervical cytology testing at the time of 6-month follow-up.
Cervical cytology testing at 12-month follow-up | 12-month follow-up
  All participants were tested for Cervical cytology testing at the time of 12-month follow-up.
Cervical cytology testing at 18-month follow-up | 18-month follow-up
  All participants were tested for Cervical cytology testing at the time of 18-month follow-up.
Cervical cytology testing at 24-month follow-up | 24-month follow-up
  All participants were tested for Cervical cytology testing at the time of 24-month follow-up.
Human Papillomavirus (HPV) genotyping tests at baseline | Baseline
  All participants underwent Human Papillomavirus (HPV) genotyping tests at baseline.
Human Papillomavirus (HPV) genotyping tests at 6-month follow-up | 6-month follow-up
  All participants underwent Human Papillomavirus (HPV) genotyping tests at 6-month follow-up.
Human Papillomavirus (HPV) genotyping tests at 12-month follow-up | 12-month follow-up
  All participants underwent Human Papillomavirus (HPV) genotyping tests at 12-month follow-up.
Human Papillomavirus (HPV) genotyping tests at 18-month follow-up | 18-month follow-up
  All participants underwent Human Papillomavirus (HPV) genotyping tests at 18-month follow-up.
Human Papillomavirus (HPV) genotyping tests at 24-month follow-up | 24-month follow-up
  All participants underwent Human Papillomavirus (HPV) genotyping tests at 24-month follow-up.

SECONDARY OUTCOMES:
16SrRNA sequencing of the vaginal secretions at baseline | Baseline
  All participants underwent vaginal secretion sequencing at baseline.
16SrRNA sequencing of the vaginal secretions at 6-month follow-up | 6-month follow-up
  All participants underwent vaginal secretion sequencing at 6-month follow-up.
16SrRNA sequencing of the vaginal secretions at 12-month follow-up | 12-month follow-up
  All participants underwent vaginal secretion sequencing at 12-month follow-up.
16SrRNA sequencing of the vaginal secretions at 18-month follow-up | 18-month follow-up
  All participants underwent vaginal secretion sequencing at 18-month follow-up.
16SrRNA sequencing of the vaginal secretions at 24-month follow-up | 24-month follow-up
  All participants underwent vaginal secretion sequencing at 24-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Binhua Dong, MD, Study Chair — Fujian Maternity and Child Health Hospital
Locations (11):
- China (11):
  - Fujian Maternity and Child Health Hospital, Fuzhou, Fujian
  - Mindong Hospital of Ningde City, Ningde, Fujian
  - Ningde Municipal Hospital of Ningde Normal University, Ningde, Fujian
  - The First Hospital of Putian City, Putian, Fujian
  - Quanzhou First Hospital Afflicated to Fujian Medical University, Quanzhou, Fujian
  - Xiamen Maternity and Child Health Hospital Affiliated to Xiamen University, Xiamen, Fujian
  - Zhangzhou affiliated Hospital of Fujian Medical University, Zhangzhou, Fujian
  - Longyan First Hospital, Longyan
  - Nanping Second Hospital, Nanjing
  - Sanming Second Hospital, Sanming
  - Shenzhen Maternity and child Healthcare Hospital, Shenzhen